CLINICAL TRIAL: NCT02163967
Title: Effect of Cranial Electrical Stimulation (CES) on Autonomic Regulation
Brief Title: Effect of CES on Parasympathetic Tone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Fisher Wallace Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: WCMC1209013001
Record Dates: First submitted 2013-02-05; First posted 2014-06-16 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: cranial electrical stimulation; CES; heart rate variability; parasympathetic; Vagal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Individual calculating heart rate and heart rate variability from ECG recordings was blind to dose of stimulation. Individual collecting side effect information was not blind to dose of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Dose sequence: Sham, Low, High (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- Sham stimulation; Day 2 -1 milliamp stimulation intensity, Day 3 - 2milliamp stimulation intensity
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)
- Dose sequence: Sham, High, Low (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- Sham stimulation; Day 2 -2 milliamp stimulation intensity, Day 3 - 1milliamp stimulation intensity
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)
- Dose sequence: Low, Sham, High (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- 1milliamp stimulation intensity; Day 2 -Sham stimulation; Day 3 - 2milliamp stimulation intensity
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)
- Dose sequence: Low, High, Sham (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- 1milliamp stimulation intensity; Day 2 - 2milliamp stimulation intensity; Day 3 - Sham stimulation
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)
- Dose sequence: High, Sham, Low (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- 2 milliamp stimulation intensity; Day 2 - Sham stimulation; Day 3 - 1 milliamp stimulation intensity
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)
- Dose sequence: High, Low, Sham (Other): Cranial Electrical Stimulation with Fisher-Wallace Stimulator (Model FW100) for 20 minutes on 3 separate days. Day 1- 2 milliamp stimulation intensity; Day 2 - 1 milliamp stimulation intensity; Day 3 - Sham stimulation
  Interventions: Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100)

INTERVENTIONS:
Device: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100) — low voltage alternating current transcranial electrical stimulation
  Other Names: Fisher-Wallace Stimulator (Model FW100)

SUMMARY:
The hypothesis is that CES stimulation will dose dependently increase parasympathetic tone. Healthy subjects will have three 20 minute sessions of CES stimulation, at three different intensities of stimulation, with each session occurring on a separate day. Effect on parasympathetic tone will determined by measuring high frequency heart rate variability before, during and after the stimulation. The Fisher Wallace Stimulator (FW100) which delivers a low dose alternating current a varying frequencies will be used for the stimulation.

DETAILED DESCRIPTION:
Healthy subjects will have three 20 minute sessions of bitemporal CES stimulation, at three different intensities of stimulation (sham, 1 milli Amp, 2 milli Amp), with each session occurring on a separate day. The Fisher Wallace Stimulator (FW100) which delivers a low dose alternating current a varying pulsed frequencies (5 Hertz, 500 Hertz, and 25000 Hertzz) will be used for the stimulation. ECG will be recorded continuously for 15 minutes before stimulation, during 20 minute stimulation and for 15 minutes following stimulation. Effect on parasympathetic tone will determined by measuring high frequency heart rate variability before, during and after the stimulation. Effect of CES of heart rate and low frequency heart rate variability will also be examined. Subject side effects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* daily psychotropic medication,
* use of beta blocker,
* pacemaker,
* other metal in body,
* history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2013-03-15 (Actual); Study Completion 2013-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Altemus, MD, Principal Investigator — Weill Medical College, Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Sequence: Sham, Low, High: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - Sham stimulation, Day 2 - 1milliamp stimulation intensity, Day 3 - 2 milliamp stimulation intensity
- Dose Sequence: Sham, High, Low: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - Sham stimulation, Day 2 - 2 milliamp stimulation intensity, Day 3 - 1 milliamp stimulation intensity
- Dose Sequence: Low, Sham, High: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - 1 milliamp stimulation intensity , Day 2 - Sham stimulation, Day 3 - 2 milliamp stimulation intensity
- Dose Sequence; Low, High, Sham: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - 1 milliamp stimulation intensity , Day 2 - 2 milliamp stimulation intensity, Day 3 - Sham stimulation
- Dose Sequence: High, Sham, Low: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - 2 milliamp stimulation intensity , Day 2 - Sham stimulation, Day 3 - 1 milliamp stimulation intensity
- Dose Sequence: High, Low, Sham: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes on 3 separate days. Day 1 - 2 milliamp stimulation intensity , Day 2 - 1 milliamp stimulation intensity, Day 3 - Sham stimulation
Period: First Intervention/ Day 1
Arm/Group | Dose Sequence: Sham, Low, High | Dose Sequence: Sham, High, Low | Dose Sequence: Low, Sham, High | Dose Sequence; Low, High, Sham | Dose Sequence: High, Sham, Low | Dose Sequence: High, Low, Sham
Started | 4 | 4 | 3 | 4 | 3 | 3
Completed | 4 | 4 | 3 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intevention/Day 2
Arm/Group | Dose Sequence: Sham, Low, High | Dose Sequence: Sham, High, Low | Dose Sequence: Low, Sham, High | Dose Sequence; Low, High, Sham | Dose Sequence: High, Sham, Low | Dose Sequence: High, Low, Sham
Started | 3 | 4 | 2 | 4 | 3 | 3
Completed | 3 | 4 | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention/Day 3
Arm/Group | Dose Sequence: Sham, Low, High | Dose Sequence: Sham, High, Low | Dose Sequence: Low, Sham, High | Dose Sequence; Low, High, Sham | Dose Sequence: High, Sham, Low | Dose Sequence: High, Low, Sham
Started | 3 | 3 | 2 | 4 | 3 | 3
Completed | 3 | 3 | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is restricted to subjects who completed all three study sessions
Groups:
- All Study Participants: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): low voltage alternating current transcranial electrical stimulation, stimulation for 20 minutes on 3 separate days. Subjects were randomized to order of stimulation dose on the 3 days.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in High Frequency Heart Rate Variability
Description: High frequency heart rate variability (HRV) will be calculated over successive 5 minute intervals from continuous ECG recordings and reported on a log scale with a minimum of 0 and a maximum of 10. Higher scores represent more heart rate variability.
Time Frame: Mean HRV is calculated for the 15 minutes of baseline, for the 20 minutes of stimulation and for the 15 minutes post stimulation
Population: 3 subjects who did not complete testing sessions at all 3 stimulation doses we not included in the final analysis
Measure: Mean (Standard Error); unit: Units on a Log Scale
Groups:
- Sham Stimulation: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): sham stimulation for 20 minutes
- Low Dose: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes at 1 milliamp stimulation dose
- High Dose: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): for 20 minutes at 2 milliamp stimulation dose
Arm/Group | Sham Stimulation | Low Dose | High Dose
Number analyzed (Participants) | 18 | 18 | 18
Units on a Log Scale
  Baseline | 5.10 (0.40) | 5.14 (0.36) | 5.00 (0.43)
  Stimulation | 5.12 (.25) | 5.36 (.23) | 5.44 (.27)
  Post Stimulation | 5.12 (.36) | 5.40 (.34) | 5.46 (.35)
Statistical Analysis 1: Comparison: Sham Stimulation vs Low Dose vs High Dose; The null hypothesis is that there is no difference in High frequency HRV after 20 minutes of stimulation or 15 minutes after cessation of stimulation at the low (1mAmp) or high (2mAmp) dose compared to sham stimulation; Test type: Other; p < .02, Regression, Linear — Mixed effects regression model, a nested (within subject) random intercept for dose, fixed effects for age, dose, time and dose x time interaction. Significance level p=.05, Bonferonni correction was used for post-hoc tests; Post-hoc comparisons using least-square means. Kenward-Roger adjustments to denominator degrees of freedom.Increase in HRV at 2Amp compared to sham

2. Secondary Outcome: Number of Subjects Reporting Light Flickering in Peripheral Vision Side Effect
Description: Subjects were asked to report any side effects of the stimulation. Of all side effects reported by subjects, only light flickering in peripheral vision was endorsed by enough subjects to allow statistical analysis
Time Frame: one hour
Population: All 21 subjects who completed at least one of the stimulation study visits are included in this analysis
Measure: Number; unit: participants
Groups:
- Sham: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100) sham stimulation for 20 minutes, once
  Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): low voltage alternating current transcranial electrical stimulation
- Low Dose: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100) 1mAmp stimulation for 20 minutes, once
  Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): low voltage alternating current transcranial electrical stimulation
- High Dose: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100) 2mAmp stimulation for 20 minutes, once
  Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): low voltage alternating current transcranial electrical stimulation
Arm/Group | Sham | Low Dose | High Dose
Number analyzed (Participants) | 20 | 19 | 18
participants | 0 | 8 | 12
Statistical Analysis 1: Comparison: Sham vs Low Dose vs High Dose; The null hypothesis is that there will be no difference in the number of side effects reported during either dose of stimulation compared to sham stimulation. Statistical differences were examined for light flickering in peripheral vision . Other side effects were reported by too few subjects to be analyzed statistically; Test type: Other; p < .001, Chi-squared

3. Secondary Outcome: Change in Heart Rate
Description: Heart rate will be calculated over successive 5 minute intervals from continuous ECG recordings. Higher scores represent faster heart rate
Time Frame: Mean heart rate is calculated for the 15 minutes of baseline, for the 20 minutes of stimulation and for the 15 minutes post stimulation
Population: 3 subjects who did not complete all 3 stimulation sessions were not included in the analysis
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Sham | Low Dose | High Dose
Number analyzed (Participants) | 18 | 18 | 18
beats per minute
  Baseline | 70.4 (1.4) | 71.8 (2.1) | 73.6 (1.8)
  Stimulation | 69.4 (1.3) | 70.1 (2.0) | 71.4 (2.1)
  Post Stimulation | 68.3 (1.2) | 69.1 (1.8) | 70.7 (1.8)
Statistical Analysis 1: Comparison: Sham vs Low Dose vs High Dose; Test type: Other; p = 0.81, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Post-hoc comparisons were made using least-square means. Kenward-Roger adjustments to denominator degrees of freedom

4. Secondary Outcome: Change in Low Frequency Heart Rate Variability
Description: Low frequency heart rate variability will be calculated over successive 5 minute intervals from continuous ECG recordings and reported on a log scale with a minimum of 0 and a maximum of 10. Higher scores represent more heart rate variability.
Time Frame: Low frequency heart rate variability is calculated for the 15 minutes of baseline, for the 20 minutes of stimulation and for the 15 minutes post stimulation
Population: 3 enrolled subjects who did not complete all 3 stimulation sessions were not included in the analysis.
Measure: Mean (Standard Error); unit: Units on a Log Scale
Arm/Group | Sham | Low Dose | High Dose
Number analyzed (Participants) | 18 | 18 | 18
Units on a Log Scale
  Baseline | 5.21 (0.21) | 5.29 (0.33) | 5.01 (0.34)
  Stimulation | 5.34 (0.21) | 5.29 (0.32) | 5.18 (0.32)
  Post-stimulation | 5.56 (0.21) | 5.43 (0.30) | 5.17 (0.29)
Statistical Analysis 1: Comparison: Sham vs Low Dose vs High Dose; Test type: Other; p = 0.47, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Post-hoc comparisons were made using least-square means. Kenward-Roger adjustments to denominator degrees of freedom

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Of the 21 subjects enrolled, 20 participated in the sham stimulation session, 19 participated in the low dose stimulation session and 18 participated in the high dose stimulation session.
Groups:
- Low Dose: Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100) 1mAmp stimulation for 20 mintues, once
  Cranial Electrical Stimulation Fisher-Wallace Stimulator (Model FW100): low voltage alternating current transcranial electrical stimulation
Arm/Group | Sham | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 1/20 | 11/19 | 12/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=20) | Low Dose (N=19) | High Dose (N=18)
light flickering (Nervous system disorders) | 0 (0) | 8 (8) | 12 (12) — flickering light in periphery of visual field during stimulation, which is not present during post-stimulation period.
itching or tingling of scalp (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3) — sense of tingling or itching at scalp contact site of electrode

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes